CLINICAL TRIAL: NCT00610194
Title: A Multi-Center Phase 1, Dose-Escalation Trial to Determine the Safety and Pharmacokinetics/Pharmacodynamics of RDEA119, A MEK Inhibitor, in Advanced Cancer Patients
Brief Title: Phase 1 Dose-escalation PK/PD Trial in Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15505; RDEA119-101 (Other: Ardea)
Record Dates: First submitted 2008-01-02; First posted 2008-02-07 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — N-(3,4-difluoro-2-(2-fluoro-4-iodophenylamino)-6-methoxyphenyl)-1-(2,3-dihydroxypropyl)cyclopropane-1-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): In the dose escalation phase, subjects will receive a single oral dose of RDEA119 on Day 1, wait 1 week, then begin a 28-day course of daily continuous dosing of RDEA119. In the expanded MTD phase, subjects will receive RDEA119 once or twice a day beginning on Day 1, and begin a 28-day course of continuous dosing at that time.
  Interventions: Drug: RDEA119

INTERVENTIONS:
Drug: RDEA119 — In the dose escalation phase, subjects will receive a single oral dose of RDEA119 on Day 1, wait 1 week, then begin a 28-day course of daily continuous dosing of RDEA119. In the expanded MTD phase, subjects will receive RDEA119 once or twice a day beginning on Day 1, and begin a 28-day course of continuous dosing at that time.

SUMMARY:
Primary Objective: To evaluate the safety of escalating oral doses of RDEA119, a MEK inhibitor, in advanced cancer patients.

Secondary Objectives:

* To describe the initial PK of different doses of RDEA119 when given once orally on Day 1 of the study
* To describe the PK of different doses of RDEA119 when given orally as continuous dosing.
* To examine the inhibition of MEK products (p-ERK), cytokine products, and other protein biomarkers
* To expand the MTD dose cohort to evaluate the safety, tolerability and PK/PD of the recommended Phase 2 dose
* To explore the presence of genotype, PD markers, cell growth and a marker of apoptosis, in paired tumor biopsy samples of patients' tumors pre-dose and during dosing in a minimum of 10 patients in the expanded cohort

ELIGIBILITY:
Inclusion Criteria: - Histological or cytological confirmed solid tumor. - Advanced metastatic or locally recurrent disease for which no proven effective therapy exists. - In the expanded MTD cohort, a minimum of 10 patients must have an accessible tumor that is amendable to biopsy (cut or needle) at the start and during the study. For patients not in the biopsy group, a block from the patient's original diagnostic biopsy/excision, if available, may be used for genotype analysis. - ECOG performance status of 0-1. - Life expectancy of > or equal to 3 months. - Acceptable hematology, clinical chemistry, and coagulation laboratory values. - Patient must be acceptable for treatment and follow up according to the Investigator. - Patent must have agreed to and signed the Informed Consent. - Patient has within normal range cardiac function as measured by echocardiogram or MUGA scan. Exclusion Criteria: - Use of investigational agents or devices within the last 28 days. - Major surgery within 30 days of start of study. - Patients with documented CNS metastasis who are not off steroids and other CNS therapies - Evidence of uncontrolled active infections. - Other serious medical or psychiatric illness. - Significant cardiac dysfunction including congestive heart failure (NYHA Class III or IV); myocardial infarction or ventricular tachyarrhythmia within the last 6 months; major conduction abnormalities unless corrected with a cardiac pacemaker; prolonged QTc >460msec. - Patients with known hypersensitivity to any of the drugs or components given in this protocol. - Pregnancy. - Women or men of childbearing potential not willing to use effective contraception, including barrier protection. - Patients with abdominal fistula, GI perforation, intra-abdominal abscess, or small bowel resection, any of which is within 6 months of study entry. - Patients with abdominal radiation resulting in chronic diarrhea. - Because RDEA119 is primarily metabolized by CYP3A4 and CYP2C19, inhibitors and inducers of these enzymes should be avoided. - Patients with known HIV infection will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-11-28 (Actual); Primary Completion 2010-11-24 (Actual); Study Completion 2012-08-01 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed as adverse and drug related events, clinical laboratory test results (hematology, chemistry, coagulation, and urinalysis), vital signs, 12-lead electrocardiograms (ECGs), and physical examination | 35 Days

SECONDARY OUTCOMES:
Pharmacokinetics and Pharmacodynamics | 35 Days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- United States (3):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - UCHSC, Aurora, Colorado
  - Roswell Park Cancer, Buffalo, New York

REFERENCES:
- [Result] Weekes CD, Von Hoff DD, Adjei AA, Leffingwell DP, Eckhardt SG, Gore L, Lewis KD, Weiss GJ, Ramanathan RK, Dy GK, Ma WW, Sheedy B, Iverson C, Miner JN, Shen Z, Yeh LT, Dubowy RL, Jeffers M, Rajagopalan P, Clendeninn NJ. Multicenter phase I trial of the mitogen-activated protein kinase 1/2 inhibitor BAY 86-9766 in patients with advanced cancer. Clin Cancer Res. 2013 Mar 1;19(5):1232-43. doi: 10.1158/1078-0432.CCR-12-3529. Epub 2013 Feb 22. PMID 23434733